CLINICAL TRIAL: NCT03538405
Title: Short-term Effect of Positioning Cushions and Harmonic Techniques on Paratonia in Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/2016/0019
Record Dates: First submitted 2018-04-17; First posted 2018-05-29 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Dementia; Paratonia
Keywords: harmonic techniques; supporting cushions; intervention
MeSH Terms: conditions — Dementia; Muscle Rigidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all participants (Experimental): All participants received the same interventions, there were no subgroups interventions: supporting cushions and harmonic techniques
  Interventions: Other: Supporting cushions; Other: Harmonic techniques

INTERVENTIONS:
Other: Supporting cushions — Cushions were placed in a way that the head and four limbs were well supported, without leaving empty space between body and cushions or mattress.
Other: Harmonic techniques — Harmonic techniques (HT) is a group of manual techniques described by Lederman (2000).The goal of this techniques in this study was to reduce the muscle tone and additionally/subsequently increase the ROM.

SUMMARY:
This study investigated the short-term effect of both harmonic techniques and supporting cushions on muscle tone, range of motion, pain and daily care activities in 22 patients with moderate to severe paratonia. The study consisted of two parts, each part was conducted during one week. In the first part of the study the short-term effect of supporting cushions was examined; in the second part of the study the additional short-term effect of harmonic techniques was investigated.

ELIGIBILITY:
Inclusion Criteria:

* dementia (confirmed in medical file)
* presence of moderate to severe paratonia (confirmed with PAI and MAS)
* proxy consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-04-24 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Change in muscle tone of biceps brachii and rectus femoris | On each measurement moment (3 or 4 times a day, 3 different days, 2 weeks for each participant)
  Change in MyotonPRO measurement of intrinsic muscle tone of left and right biceps brachii and left and right rectus femoris
Change in maximal extension of elbow and knee | On each measurement moment (3 or 4 times a day, 3 different days, 2 weeks for each participant)
  Change in goniometric measurement of maximal elbow and knee extension
Change in pain | On each measurement moment (3 or 4 times a day, 3 different days, 2 weeks for each participant)
  Change in PACSLAC-D score (PACSLAC-D is a Dutch adaptation of the Pain Assessment Checklist for Seniors with Limited Ability to Communicate): observation scale of pain during morning care. Scores range from 0 to 24, indicating the presence of various pain expressions. Higher scores indicate more pain.
Comparison of pain during morning care | rated after morning care, daily during 2 weeks for each participant (control week and intervention week)
  Comparison of PACSLAC-D scores during control week and harmonics week.PACSLAC-D is a Dutch adaptation of the Pain Assessment Checklist for Seniors with Limited Ability to Communicate: observation scale of pain during morning care. Scores range from 0 to 24, indicating the presence of various pain expressions. Higher scores indicate more pain.
Comparison of comfort during morning care | rated after morning care, daily during 2 weeks for each participant (control week and intervention week)
  Comparison of score on comfort questionnaire 4 questions regarding comfort of morning care (both for caregiver as estimated for patient) between control week and harmonics week, as rated with a visual analogue scale (0-10, interpretation dependent on the question)

OTHER OUTCOMES:
diagnosis of paratonia | for inclusion
  Paratonia Assessment Instrument, resistance against passive movements of the four limbs is evaluated (Hobbelen 2008)
paratonia severity | for inclusion
  Rating of paratonia severity by means of the Modified Ashworth Scale (MAS). Resistance against passive movement of the limbs is rated. Scores: 0: Normal tone, passive movement no problem; 1: Mild paratonia, slight resistance in passive movement; 2: Moderate paratonia, enhanced resistance in passive movement; 3: Severe paratonia, severe resistance in passive movement; 4: Very severe paratonia, passive movement (almost) impossible. Participants with moderate to severe paratonia were included in this study, defined as presence of a MAS score of ≥2 in at least one limb

CONTACTS AND LOCATIONS:
Locations (1):
- Vakgroep Revaki - Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided